CLINICAL TRIAL: NCT03793335
Title: Individually Tailored Strategies for the Precision Prevention of Gastric Cancer and Colorectal Cancer in the Community
Status: Enrolling by invitation | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201811034RINB
Record Dates: First submitted 2019-01-02; First posted 2019-01-04 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Gastric Cancer; Colorectal Cancer
MeSH Terms: conditions — Stomach Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gastric cancer prevention: This prospective study consists of 40,000 participants; after randomization, each arm has 20,000 participants. Arm 1: participants receive H. pylori stool antigen test; Arm 2: participants receive the combination of H. pylori stool antigen test and serum pepsinogen test.
- Colorectal cancer prevention: This prospective study consists of 40,000 participants; after randomization; each arm has 20,000 participants. Arm 1: participants with positive fecal immunochemical test (FIT) receive routine referral confirmatory diagnosis approach; Arm 2: participants with positive FIT receive routine referral confirmatory diagnosis approach and participants with high FIT results receive additional aggressive referral confirmatory diagnosis approach.

SUMMARY:
Gastric cancer is a global health threat. Helicobacter pylori is now recognized as the main risk factor that initiates this process; hence, H. pylori eradication has been considered the most effective method to ameliorate the burden of gastric cancer. Serum pepsinogen levels reveal the current atrophy of the stomach and predict gastric cancer risk. A risk prediction model with the combination of H. pylori infection and serum pepsinogen level could identify the highest-risk gastric cancer patients.

Colorectal cancers (CRC) rank second and third as the leading causes of cancer-related death in men and women, respectively. For CRC prevention, a two-stage approach using the fecal immunochemical test (FIT) is popular; besides, the FIT levels may serve as a guide for priority setting in prompting residents to undergo colonoscopy. Therefore, the effectiveness and utility of aggressive referral confirmatory diagnosis protocol in a colorectal cancer screening program for those with high FIT levels urgently need to evaluate.

DETAILED DESCRIPTION:
Gastric cancer is a global health threat and contributes to more than 720,000 deaths per year. In the absence of early detection, gastric cancer is associated with a high fatality rate-the 5-year survival rate for patients with locally advanced disease is only about 40% despite aggressive treatment. Carcinogenesis in gastric cancer follows a multistage process (i.e., Correa's model) that develops from chronic active gastritis to atrophic gastritis, intestinal metaplasia, dysplasia, and finally to carcinoma. Helicobacter pylori is now recognized as the main risk factor that initiates this process. An estimated 89% of non-cardiac cancers can be prevented if H. pylori can be eradicated from the population of interest; hence, H. pylori eradication has been considered the most effective method to ameliorate the burden of gastric cancer. However, in the setting of mass screening, irreversible damage may already have occurred after patients have harbored H. pylori infection for decades before they undergo screening and treatment for H. pylori. This observation has been supported by a recent meta-analysis based on 8 randomized controlled trials and 16 cohort studies that investigated the magnitude of the benefit from eradication therapy; on average, only a 50% reduction of gastric cancer risk was shown. Altered levels of serum pepsinogens, which are mainly produced by the chief cells of the fundic glands of the stomach, reflect the atrophic status (ie, gland loss) of gastric mucosa. Serum pepsinogen levels not only reveal the past infection status or current atrophy of the stomach, respectively, but have also been shown to be predictive of gastric cancer risk. Therefore, to completely eliminate the burden of gastric cancer, physicians urgently need a risk prediction model with the combination of H. pylori infection and serum pepsinogen level to identify the highest-risk patients for endoscopic examination in the context of limited resources.

Colorectal cancers (CRC) rank second and third as the leading causes of cancer-related death in men and women, respectively, in the world. To reduce the burden of CRC, colonoscopy is the most effective method and can reduce the risk of new-onset CRCs by the removal of adenomatous polyps and can improve CRC survival by the detection of pre-symptomatic malignancies. In addition to primary screening colonoscopy, a two-stage approach using the fecal immunochemical test (FIT) is increasingly popular because of its ability to identify patients with the highest risk of CRC; in this manner, limited colonoscopist resources can be efficiently allocated. Although colonoscopy is associated with a statistically significant reduction in mortality rates for CRC through the detection of early-stage cancers, the FIT levels may serve as a guide for priority setting in prompting residents to undergo colonoscopy. Besides, the prevalence of any CRC and advanced-stage CRC is associated with delays in follow-up colonoscopies for patients with positive results from a FIT. Therefore, the effectiveness and utility of aggressive referral confirmatory diagnosis protocol in a colorectal cancer screening program for those with high FIT levels urgently need to evaluate.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 50-75 years
2. Confirmed non-gastric cancer/colorectal cancer healthy participant
3. Mentally competent to be able to understand the consent form
4. Able to communicate with study staff for individuals
5. Agree to link the screening data to National Cancer Registry

Exclusion Criteria:

1. Confirmed gastric cancer/colorectal cancer healthy participant
2. Status post gastrectomy

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A community-based mass screening for gastric cancer and colorectal cancer is designed and targeted at community residents aged 50-75 years in Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2019-04-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Gastric cancer prevention | Up to 10 years, the gastric cancer incidence per 100,000 person-years is calculated by the person-years of follow-up.
  To assess the combination of H. pylori stool antigen test and serum pepsinogen test as a joint predictor of gastric cancer risk
Colorectal cancer prevention | Up to 10 years, the colorectal cancer incidence per 100,000 person-years is calculated by the person-years of follow-up.
  To assess the effectiveness/utility of aggressive referral confirmatory diagnosis protocol in a colorectal cancer screening program

CONTACTS AND LOCATIONS:
Overall Officials: TSUNG-HSIEN CHIANG, MD, MSc, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
No individual participant data could be shared.